CLINICAL TRIAL: NCT01749449
Title: Increased Protein Intake and Meal Frequency Reduces Abdominal Fat and Increases Postprandial Thermogenesis During Energy Balance and Energy Deficit
Brief Title: Increased Dietary Protein and Meal Frequency Reduces Total and Abdominal Body Fat During Weight Maintenance and Weight Loss
Acronym: 3v6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3v6-021904
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2007-01

CONDITIONS: Obesity
Keywords: high protein; high carbohydrate; meal frequency; abdominal body fat; postprandial thermogenesis
MeSH Terms: conditions — Obesity | interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High protein 3 meals/day (Experimental): 35% protein intake eaten as 3 meals per day
  Interventions: Other: protein and meal frequency
- High carbohydrate consumed 3 meals/day (Experimental): High carbohydrate 3 meals/day
  Interventions: Other: protein and meal frequency
- High protein consumed 6 meals/day (Experimental): 35% protein 6 meals/day
  Interventions: Other: protein and meal frequency

INTERVENTIONS:
Other: protein and meal frequency — comparison of different levels of protein intake and meal frequency on body composition in obese adults

SUMMARY:
The purpose of the current study was to examine the impact of macronutrient intake (PRO, 15% vs. 35%) and meal frequency (3 vs. 6 meals/day) on body composition, postprandial thermogenesis and plasma adipokines before and after 28days each of EB (28days) and ED (25%; 28days) in overweight individuals. We hypothesize that HP will elicit more favorable body composition, thermogenic, and cardiometabolic changes than HC intakes and the magnitude of change will be greatest in those consuming HP meals more frequently.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years old,
* overweight or obese but otherwise in good health

Exclusion Criteria:

* cardiovascular disease,
* cancer,
* HTN,
* type I or II DM,
* food allergies

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2006-05 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
body composition | 2 months
  DXA was used to quantify changes in body composition over the 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Arciero, PhD, Principal Investigator — Skidmore College
Locations (1):
- Skidmore College, Saratoga Springs, New York, United States